CLINICAL TRIAL: NCT05735470
Title: An Exploratory Clinical Trial to Evaluate the Efficacy and Safety of a Novel Antibacterial Bone Traction Needle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021 0873
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Wound Infection
Keywords: external fixation, implant
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibacterial bone traction needle (Experimental): The bone traction needle with an antibacterial coating.
  Interventions: Device: antibacterial bone traction needles
- bone traction needle (No Intervention): The bone traction needle without an antibacterial coating.

INTERVENTIONS:
Device: antibacterial bone traction needles — Whether to use bone traction needles containing antibacterial coatings
  Arms: Antibacterial bone traction needle

SUMMARY:
The goal of this clinical trial is to test in wound infection. The main question it aims to answer is: Whether this antibacterial bone traction needle is safe and has a good effect on wound infection. Participants will be implanted with an antibacterial bone traction needles and the infection grade of wound after surgery will be observed. If there is a comparison group: Researchers will compare the control group without antibacterial ability to see if the experimental group Can effectively inhibit wound infection.

ELIGIBILITY:
Inclusion Criteria:

1. Limb fractures, infections, defects and deformities caused by various congenital or acquired factors, such as multiple fractures of tibia and fibula, infectious bone defects of tibia, knee varus, horseshoe varus foot, etc.;
2. The subject understands the significance of this project, voluntarily acts as the subject and signs the informed consent.

Exclusion Criteria:

1. The subjects are pregnant or lactating women;
2. Pathological fractures (such as primary or metastatic tumors);
3. The patient is allergic to iodine and its compounds;
4. The patient is allergic to metal implants;
5. Patients with coagulopathy (such as hemophilia, vitamin K deficiency, severe liver disease, etc.);
6. The patient had participated in other clinical trials in the past 3 months;
7. The patient had contraindications to anesthesia and surgery;
8. The patient is currently receiving chemotherapy or radiotherapy, systemic corticosteroid use (continuous use for more than 3 months);
9. The patient had poor compliance and was judged by the researchers to be unable to complete the experiment according to the research plan, such as alcohol addiction, drug abuse, schizophrenia, dementia, and did not provide consent for voluntary participation in the clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Wound healing grading | 3 months
  The wound healing grading is evaluated by combining the wound healing grading, Sims grading and VAS grading

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoming Ye, Doctor, Study Chair — 2' affiliated Hospital, Schoolc of Medcine, Zhejiang University, China
Locations (1):
- Zhaoming Ye, Hangzhou, Zhejiang, China